CLINICAL TRIAL: NCT04624243
Title: A Phase 2B Randomized, Double-Blind, Placebo- and Active-Controlled Trial of the Efficacy and Safety of MK-8189 in Participants Experiencing an Acute Episode of Schizophrenia
Brief Title: Efficacy and Safety of MK-8189 in Participants With an Acute Episode of Schizophrenia (MK-8189-008)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 8189-008; MK-8189-008 (Other: Merck Protocol Number); jRCT2071200096 (Registry Identifier: jRCT); 2020-000094-24 (EudraCT Number)
Record Dates: First submitted 2020-11-05; First posted 2020-11-10 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — MK-8189; Risperidone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- MK-8189 8 mg (Experimental): Participants received MK-8189 8 mg QD from Weeks 1 to 12, with 2 weeks of follow-up
  Interventions: Drug: MK-8189; Drug: Placebo to risperidone
- MK-8189 16 mg (Experimental): Participants received MK-8189 16 mg QD from Weeks 1 to 12, with 2 weeks of follow-up.
  Interventions: Drug: MK-8189; Drug: Placebo to risperidone
- MK-8189 24 mg (Experimental): Participants received MK-8189 24 mg QD from Weeks 1 to 12, with 2 weeks of follow-up.
  Interventions: Drug: MK-8189; Drug: Placebo to risperidone
- Risperidone 6 mg (Active Comparator): Participants will be treated for a total of 12 weeks. Participants will receive risperidone 6 mg QD in the acute treatment period from Week 1-6 followed by risperidone 6 mg QD in the extension treatment period from Week 7-12.
  Interventions: Drug: Risperidone; Drug: Placebo to MK-8189
- Placebo and MK-8189 24 mg (Experimental): Participants received placebo QD from Weeks 1 to 6 and MK-8189 24 mg from Weeks 7 to 12, with 2 weeks of follow-up.
  Interventions: Drug: MK-8189; Drug: Placebo to MK-8189; Drug: Placebo to risperidone

INTERVENTIONS:
Drug: MK-8189 — MK-8189 administered QD at a dose of 8 mg, 16 mg, or 24 mg via oral tablet.
  Arms: MK-8189 16 mg; MK-8189 24 mg; MK-8189 8 mg; Placebo and MK-8189 24 mg
Drug: Risperidone — Risperidone administered QD at a dose of 6 mg via oral capsule.
  Arms: Risperidone 6 mg
Drug: Placebo to MK-8189 — MK-8189-matching placebo administered QD via oral tablet.
  Arms: Placebo and MK-8189 24 mg; Risperidone 6 mg
Drug: Placebo to risperidone — Risperidone-matching placebo administered QD via oral capsule.
  Arms: MK-8189 16 mg; MK-8189 24 mg; MK-8189 8 mg; Placebo and MK-8189 24 mg

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of MK-8189 at a range of doses (8 mg, 16 mg, and 24 mg once daily [QD]) in adult participants who have an acute episode of schizophrenia according to Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM-5) criteria. The primary hypotheses were the following: (1) that MK-8189 24 mg is superior to placebo in reducing the Week 6 mean change from baseline in Positive and Negative Syndrome Scale (PANSS) total score, and (2) that MK-8189 16 mg is superior to placebo in reducing the Week 6 mean change from baseline in PANSS total score.

With Amendment 4, enrollment was changed to approximately 500 participants with removal of the MK-8189 8 mg treatment arm. Participants enrolled before Amendment 4 who were assigned to MK-8189 8 mg QD remained on that dose regimen per protocol.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include, but are not limited to the following:

* Meet the diagnostic criteria for schizophrenia according to the DSM-5
* Have an illness duration for schizophrenia of at least 1 year
* Be confirmed to be experiencing an acute episode of schizophrenia as evidenced by ALL of the following: (a) onset of the current acute episode is ≤6 weeks before screening (b) current symptoms represent a marked and substantial worsening compared with the participant's usual symptomatic state prior to the current acute episode, and are associated with diminished functional ability (c) in need of increased psychiatric attention to treat worsening acute episode symptoms
* Have a CGI-S score of ≥4 (moderately ill) at screening and baseline
* Have an identified responsible person referred to as the "external contact person" who has agreed to provide information about the participant's location if needed during outpatient portion of the study. The site personnel must consider this identified responsible person a reliable contact person, and the contact person must have regular contact with the participant (defined at screening as direct contact no fewer than 3 times per week), and with the expectation that this frequency of contact would continue (either in person or via other contact method), throughout duration of the study, including the follow-up period)

Exclusion Criteria:

The main exclusion criteria include, but are not limited to the following:

* Has a primary current diagnosis other than schizophrenia or a comorbid diagnosis that is primarily responsible for the current symptoms and functional impairment
* Meets criteria for moderate to severe substance use disorder within past 6 months prior to screening (excluding those related to caffeine or nicotine)
* Has a known history of the following: (a) borderline personality disorder, anti-social personality disorder, or bipolar disorder (b) traumatic brain injury causing ongoing cognitive difficulties, Alzheimer's Disease, or another form of dementia, or any chronic organic disease of the central nervous system (c) intellectual disability of a severity that would impact ability to participate in the study
* Has a current diagnosis of a psychotic disorder other than schizophrenia or a behavioral disturbance thought to be due to substance abuse
* Is or was under involuntary commitment for the acute episode, because the participant is considered a danger to themselves or others
* Has a history of treatment resistance exhibited by any of the following: (a) no or minimal response to at least 2 periods of treatment lasting 6 weeks or longer, with antipsychotic agents at the maximally tolerated dose. Participants who have responded to antipsychotics only when paired with clozapine are considered treatment-resistant (b) history of electroconvulsive therapy (ECT) treatment for treatment-resistant schizophrenia within the past 6 months (c) past or current use of clozapine as single or adjunctive therapy for schizophrenia within the past 3 months
* Is currently participating in or has participated in another clinical study and received an experimental or investigational drug agent within 3 months prior to screening visit of this current study and has participated in no more than 2 studies in the past 2 years

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 499 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (121):
- United States (35):
  - Pillar Clinical Research ( Site 1047), Bentonville, Arkansas
  - Woodland International Research Group, LLC ( Site 1002), Little Rock, Arkansas
  - Woodland Research Northwest, LLC ( Site 1036), Rogers, Arkansas
  - CITRIALS ( Site 1010), Bellflower, California
  - ProScience Research Group ( Site 1046), Culver City, California
  - Collaborative Neuroscience Research, LLC ( Site 1041), Garden Grove, California
  - Behavioral Research Specialists, LLC ( Site 1032), Glendale, California
  - CITRIALS ( Site 1016), Riverside, California
  - Artemis Institute for Clinical Research ( Site 1019), San Diego, California
  - California Neuropsychopharmacology Clinical Research Institute, LLC (CNRI-San Diego, LLC) ( Site 103, San Diego, California
  - Schuster Medical Research Institute ( Site 1023), Sherman Oaks, California
  - Behavioral Clinical Research ( Site 1058), Hollywood, Florida
  - Research Centers of America ( Hollywood )-Central Nervous System (CNS) ( Site 1065), Hollywood, Florida
  - Premier Clinical Research Institute ( Site 1049), Miami, Florida
  - Behavioral Clinical Research , Inc ( Site 1013), Miami Lakes, Florida
  - Fort Lauderdale Behavioral Health Center ( Site 1028), Oakland Park, Florida
  - Health Synergy Clinical Research ( Site 1051), Stuart, Florida
  - Atlanta Center For Medical Research ( Site 1022), Atlanta, Georgia
  - CenExel iResearch, LLC ( Site 1039), Decatur, Georgia
  - Ascension Saint Elizabeth ( Site 1000), Chicago, Illinois
  - Uptown Research Institute ( Site 1052), Chicago, Illinois
  - Pillar Clinical Research, LLC ( Site 1038), Chicago, Illinois
  - Benchmark Research ( Site 1054), Shreveport, Louisiana
  - CBH Health ( Site 1044), Gaithersburg, Maryland
  - Massachusetts General Hospital ( Site 1035), Boston, Massachusetts
  - Arch Clinical Trials ( Site 1048), St Louis, Missouri
  - Altea Research Institute ( Site 1012), Las Vegas, Nevada
  - Hassman Research Institute Marlton Site ( Site 1040), Marlton, New Jersey
  - Richmond Behavioral Associates ( Site 1064), Staten Island, New York
  - New Hope Clinical Research ( Site 1050), Charlotte, North Carolina
  - Midwest Clinical Research ( Site 1059), Dayton, Ohio
  - Midwest Clinical Research Center ( Site 1033), Dayton, Ohio
  - Neuro-Behavioral Clinical Research ( Site 1055), North Canton, Ohio
  - Community Clinical Research ( Site 1057), Austin, Texas
  - Pillar Clinical Research, LLC ( Site 1004), Richardson, Texas
- Bulgaria (6):
  - State Psychiatric Hospital "Sv. Ivan Rilski", Novi Iskar ( Site 3001), Novi Iskar, Sofia
  - Mental Health Center Prof. Dr. Ivan Temkov - Burgas EOOD ( Site 3002), Burgas
  - State Psychiatric Hospital - Kardzhali ( Site 3005), Kardzhali
  - Mental Health Center - Ruse, EOOD ( Site 3003), Rousse
  - Center for Mental Health Prof. Nikola Shipkovenski Ltd ( Site 3000), Sofia
  - Mental Health Center - Veliko Tarnovo ( Site 3006), Veliko Tarnovo
- Croatia (4):
  - Klinika za psihijatriju Vrapce ( Site 4000), Zagreb, City of Zagreb
  - Klinika za psihijatriju Vrapce ( Site 4001), Zagreb, City of Zagreb
  - Klinicki bolnicki centar Rijeka ( Site 4005), Rijeka, Primorje-Gorski Kotar County
  - Klinika za psihijatriju Sveti Ivan ( Site 4003), Zagreb, Zagreb County
- Japan (22):
  - Seishinkai Okehazama Hospital Fujita Kokoro Care Center ( Site 2011), Toyoake, Aichi-ken
  - Kohnodai Hospital, National Center for Global Health and Medicine ( Site 2005), Ichikawa, Chiba
  - Wakato Hospital ( Site 2031), Kitakyushu, Fukuoka
  - Shiranui Hospital ( Site 2043), Omuta, Fukuoka
  - Seimou Hospital ( Site 2004), Tomioka, Gunma
  - Soushu Hospital ( Site 2008), Atsugi, Kanagawa
  - Tanzawa Hospital ( Site 2037), Hadano, Kanagawa
  - Kanagawa Psychiatric Center ( Site 2035), Yokohama, Kanagawa
  - Komoro Kogen Hospital ( Site 2046), Komoro, Nagano
  - National Hospital Organization Ryukyu Hospital ( Site 2019), Kunigamigun, Okinawa
  - Amekudai Hospital ( Site 2020), Naha, Okinawa
  - National Hospital Organization Hizen Psychiatric Medical Center ( Site 2017), Kanzaki-gun, Saga-ken
  - Rainbow and Sea Hospital ( Site 2016), Karatsu, Saga-ken
  - Ongata Hospital ( Site 2007), Hachiōji, Tokyo
  - Nishigahara Hospital ( Site 2042), Kita-ku, Tokyo
  - National Center of Neurology and Psychiatry ( Site 2023), Kodaira, Tokyo
  - Chiba University Hospital ( Site 2024), Chiba
  - Inokuchi Noma Hospital ( Site 2030), Fukuoka
  - Kuramitsu Hospital ( Site 2014), Fukuoka
  - Yuge Hospital ( Site 2018), Kumamoto
  - Seijin Hospital ( Site 2026), Tokyo
  - Narimasu Kosei Hospital ( Site 2006), Tokyo
- Latvia (2):
  - Daugavpils Psihoneirologiska Slimnica ( Site 8005), Daugavpils
  - Piejuras Slimnica Psihiatriska Klinika ( Site 8001), Liepāja
- Poland (5):
  - Centrum Medyczne HCP ( Site 0913), Poznan, Greater Poland Voivodeship
  - Klinika Psychiatryczna Wydzialu Nauki o Zdrowiu WUM ( Site 0900), Pruszków, Masovian Voivodeship
  - Samodzielny Wojewódzki Zespół Publicznych Zakładów Psychiatrycznej Opieki Zdrowotnej w Warszawie ( S, Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne ( Site 0902), Gdansk, Pomeranian Voivodeship
  - Specjal. Psychiatryczny ZOZ w Lodzi, Szpital im. Babinskiego ( Site 0905), Lodz, Łódź Voivodeship
- Romania (6):
  - Prof. Dr. Alexandru Obregia Psychiatry Hospital ( Site 0815), Bucharest, București
  - Prof. Dr. Alexandru Obregia Psychiatry Hospital ( Site 0816), Bucharest, București
  - Prof. Dr. Alexandru Obregia Psychiatry Hospital ( Site 0817), Bucharest, București
  - Prof. Dr. Alexandru Obregia Psychiatry Hospital ( Site 0818), Bucharest, București
  - Institutul de Psihiatrie Socola ( Site 0810), Iași, Iaşi
  - Institutul de Psihiatrie Socola ( Site 0814), Iași, Iaşi
- Russia (14):
  - Arkhangelsk Regional Psychiatric Clinical Hospital ( Site 6020), Arkhangelsk, Arkhangelskaya oblast
  - SGHI Leningrad Region Psyconeurology Dispensary ( Site 6017), Leningrad Region, Leningradskaya Oblast'
  - Lipetsk Regional Psychoneurology Hospital ( Site 6021), Lipetsk, Lipetsk Oblast
  - Moscow Scientific Research Institute for Psychiatry ( Site 6013), Moscow, Moscow
  - Psychiatric Clinical Hospital 4 named after PB Gannushkin ( Site 6016), Moscow, Moscow
  - Psychiatric Clinical Hospital 4 named after PB Gannushkin-Psychiatric department 4 ( Site 6023), Moscow, Moscow
  - Central Moscow Regional Clinical Psychiatric Hospital ( Site 6018), Moscow, Moscow
  - Bekhterev Research Institute for Psychoneurology ( Site 6008), Saint Petersburg, Sankt-Peterburg
  - SPb City Psychiatric Hospital #3 na II Skvortsov-Stepanov ( Site 6000), Saint Petersburg, Sankt-Peterburg
  - SPb City Psychiatric Hospital #3 na II Skvortsov-Stepanov ( Site 6001), Saint Petersburg, Sankt-Peterburg
  - SPb City Psychiatric Hospital #3 na II Skvortsov-Stepanov ( Site 6002), Saint Petersburg, Sankt-Peterburg
  - Stavropol Region Psychiatric Hospital #2 ( Site 6005), Stavropol, Stavropol Kray
  - Federal State Scientific Institution Research Institute of Mental Health ( Site 6014), Tomsk, Tomsk Oblast
  - Yaroslavl Regional Clinical Psychiatry Hospital ( Site 6022), Yaroslavl, Yaroslavl Oblast
- Serbia (9):
  - Clinical Center of Serbia ( Site 5101), Belgrade, Beograd
  - Clinical Center of Serbia ( Site 5107), Belgrade, Beograd
  - Institut za mentalno zdravlje ( Site 5105), Belgrade, Beograd
  - University Clinical Hospital Center "Dr. Dragisa Misovic - Dedinje" ( Site 5104), Belgrade, Beograd
  - Clinical Center Kragujevac ( Site 5100), Kragujevac, Sumadijski Okrug
  - Clinical Center Kragujevac ( Site 5102), Kragujevac, Sumadijski Okrug
  - Clinical Center Kragujevac ( Site 5106), Kragujevac, Sumadijski Okrug
  - Special Hospital for Psychiatric Diseases Kovin ( Site 5108), Kovin, Vojvodina
  - Special Hospital for Psychiatric Diseases Kovin ( Site 5109), Kovin, Vojvodina
- South Korea (3):
  - Inje University Busan Paik Hospital ( Site 0604), Busan, Pusan-Kwangyokshi
  - Kyungpook National University Hospital ( Site 0601), Daegu, Taegu-Kwangyokshi
  - Seoul National University Hospital ( Site 0600), Seoul
- Taiwan (5):
  - China Medical University Hospital ( Site 9006), Taichung
  - National Taiwan University Hospital ( Site 9001), Taipei
  - Taipei City Hospital, Songde Branch ( Site 9004), Taipei
  - Taipei Veterans General Hospital ( Site 9000), Taipei
  - Chang Gung Memorial Hospital - Linkou Branch ( Site 9002), Taoyuan District
- Ukraine (10):
  - CNE Cherkasy reg. psychiatric hospital of Cherkasy regional council ( Site 7009), Smila, Cherkasy Oblast
  - Dnepropetrovsk Regional Clinical Hospital Mechnikov-Regional Centre of Psychosomatic Disorders base, Dnipro, Dnipropetrovsk Oblast
  - CNE "Precarpathian Regional Clinical Center of Mental Health of Ivano-Frankivsk Regional Council"" (, Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - CNE of Kharkiv Reg. Council Reg. Clinical Psychiatric Hospital Nub 3 ( Site 7012), Kharkiv, Kharkivs’ka Oblast’
  - Institute of Neurology,Psychiatry and Narcology AMS Ukraine ( Site 7011), Kharkiv, Kharkivs’ka Oblast’
  - CNE. Kherson Regional Psychiatric Hospital ( Site 7004), Kherson, Kherson Oblast
  - Kyiv City Psychoneurological Hospital 2 ( Site 7008), Kyiv, Kyivska Oblast
  - CNE Clinical Hospital PSYCHIATRY of executive body of Kyiv City Council -Kyiv City State Admin ( Sit, Kyiv, Kyivska Oblast
  - MNE of KRC-Regional psychiatric and narcological medical association ( Site 7005), Kyiv, Kyivska Oblast
  - CNE "Vinnytsia Regional Clinical Psycho-neurological hospita-Mixed (men and women) department #2 ( S, Vinnytsia, Vinnytsia Oblast

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26833&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled and randomized at 75 study sites in 11 countries.
Pre-assignment Details: Randomization into the MK-8189 8 mg arm ceased as of Amendment 4.
Groups:
- MK-8189 8 mg: Participants received MK-8189 8 mg once daily (QD) from Weeks 1 to 12, with 2 weeks of follow-up.
- Risperidone 6 mg: Participants received risperidone 6 mg QD from Weeks 1 to 12, with 2 weeks of follow-up.
Period: Overall Study
Arm/Group | MK-8189 8 mg | MK-8189 16 mg | MK-8189 24 mg | Risperidone 6 mg | Placebo and MK-8189 24 mg
Started | 41 | 132 | 132 | 65 | 129
Completed | 14 | 64 | 61 | 37 | 70
Not Completed | 27 | 68 | 71 | 28 | 59
Not completed — Death | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 3 | 7 | 1 | 3
Not completed — Physician Decision | 3 | 8 | 15 | 2 | 11
Not completed — Withdrawal by Subject | 19 | 44 | 40 | 21 | 39
Not completed — Miscellaneous | 3 | 12 | 9 | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-8189 8 mg | MK-8189 16 mg | MK-8189 24 mg | Risperidone 6 mg | Placebo and MK-8189 24 mg | Total
Number analyzed (Participants) | 41 | 132 | 132 | 65 | 129 | 499
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.7 (8.9) | 39.4 (9.0) | 36.9 (9.2) | 38.5 (9.6) | 40.2 (9.1) | 38.5 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 46 | 42 | 25 | 42 | 167
  Male | 29 | 86 | 90 | 40 | 87 | 332
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 14 | 10 | 4 | 11 | 40
  Not Hispanic or Latino | 40 | 117 | 121 | 61 | 118 | 457
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 3 | 2 | 1 | 4 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 18 | 59 | 59 | 29 | 57 | 222
  White | 20 | 68 | 70 | 34 | 66 | 258
  More than one race | 1 | 1 | 1 | 1 | 2 | 6
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at Week 6
Description: The PANSS assesses the severity of schizophrenia symptoms through a 30-item clinician-rated inventory organized into a positive subscale (7 items), a negative subscale (7 items) and a general psychopathology subscale (16 items). For each item, symptoms are rated on a 7-point scale from 1 (absent) to 7 (extreme). The PANSS total score for each participant was calculated as the sum of the rating assigned to each of the 30 PANSS items, and ranges from 30 (lowest total score) to 210 (highest total score). Higher and lower change scores reflect symptom worsening and improvement, respectively. Risperidone and placebo were active and inactive controls, respectively.
Time Frame: Baseline and Week 6
Population: All participants who receive ≥1 dose of MK-8189 (16 mg or 24 mg), risperidone, or placebo, and have both a baseline measurement and ≥1 valid post-baseline assessment, are included. Per protocol, the effect of the 8 mg dose was not assessed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | MK-8189 8 mg | MK-8189 16 mg | MK-8189 24 mg | Risperidone 6 mg | Placebo and MK-8189 24 mg
Number analyzed (Participants) | 0 | 85 | 68 | 42 | 91
Score on a scale |  | -20.7 [-24.1 to -17.3] | -18.5 [-22.1 to -15.0] | -24.0 [-28.8 to -19.2] | -17.8 [-21.2 to -14.5]
Statistical Analysis 1: Comparison: MK-8189 16 mg vs Placebo and MK-8189 24 mg; Test type: Superiority — It was hypothesized that MK-8189 16 mg is superior to placebo in reducing Week 6 PANSS change from baseline; p = 0.241, ANCOVA; LS Mean Difference = -2.8, 97.5% CI 2-sided [-8.3 to 2.6]
Statistical Analysis 2: Comparison: MK-8189 24 mg vs Placebo and MK-8189 24 mg; Test type: Superiority — It was hypothesized that MK-8189 24 mg is superior to placebo in reducing Week 6 PANSS change from baseline; p = 0.784, ANCOVA; LS Mean Difference = -0.7, 97.5% CI 2-sided [-6.3 to 4.9]

2. Primary Outcome: Number of Participants Who Experience One or More Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporarily associated with the use of study intervention, whether or not considered related to the study intervention. Per protocol, events were assessed for the first 6 weeks of treatment.
Time Frame: Up to Week 6
Population: All participants who received ≥1 dose of study intervention are included.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-8189 8 mg | MK-8189 16 mg | MK-8189 24 mg | Risperidone 6 mg | Placebo and MK-8189 24 mg
Number analyzed (Participants) | 41 | 132 | 132 | 65 | 129
Participants | 29 | 85 | 94 | 31 | 70

3. Secondary Outcome: Change From Baseline in PANSS Positive Subscale (PSS) Score at Week 6
Description: The PANSS Positive Subscale (PSS) assesses the severity of schizophrenia symptoms. The PANSS PSS score was calculated as the sum of the rating assigned to each of the 7 PSS items and ranges from 7 (lowest total score) to 49 (highest total score). Higher and lower change scores reflect symptom worsening and improvement, respectively. Risperidone and placebo were active and inactive controls, respectively.
Time Frame: Baseline and Week 6
Population: All participants who received ≥1 dose of MK-8189 (16 mg or 24 mg), risperidone, or placebo, and have both a baseline measurement and ≥1 valid post-baseline assessment, are included. Per protocol, the effect of the 8 mg dose was not assessed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | MK-8189 8 mg | MK-8189 16 mg | MK-8189 24 mg | Risperidone 6 mg | Placebo and MK-8189 24 mg
Number analyzed (Participants) | 0 | 85 | 68 | 42 | 91
Score on a scale |  | -7.1 [-8.2 to -6.0] | -7.2 [-8.3 to -6.0] | -7.7 [-9.3 to -6.1] | -5.8 [-6.9 to -4.7]
Statistical Analysis 1: Comparison: MK-8189 16 mg vs Placebo and MK-8189 24 mg; Test type: Superiority — It was hypothesized that MK-8189 16 mg is superior to placebo in reducing Week 6 PANSS PSS change from baseline; p = 0.096, ANCOVA; LS Mean Difference = -1.3, 97.5% CI 2-sided [-3.1 to 0.5]
Statistical Analysis 2: Comparison: MK-8189 24 mg vs Placebo and MK-8189 24 mg; Test type: Superiority — It was hypothesized that MK-8189 24 mg is superior to placebo in reducing Week 6 PANSS PSS change from baseline; p = 0.094, ANCOVA; LS Mean Difference = -1.4, 97.5% CI 2-sided [-3.2 to 0.5]

4. Secondary Outcome: Change From Baseline in Clinical Global Impression-Severity of Illness (CGI-S) Score at Week 6
Description: The CGI-S is a single item 7-point clinician rated scale for assessing the global severity of the participant's illness. CGI-S scores range from 1 (participant normal, not ill) to 7 (participant extremely ill); higher and lower change from baseline scores indicate symptom worsening and improvement, respectively. Risperidone and placebo were active and inactive controls, respectively.
Time Frame: Baseline and Week 6
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | MK-8189 8 mg | MK-8189 16 mg | MK-8189 24 mg | Risperidone 6 mg | Placebo and MK-8189 24 mg
Number analyzed (Participants) | 0 | 83 | 68 | 42 | 88
Score on a scale |  | -1.1 [-1.3 to -0.9] | -1.0 [-1.2 to -0.8] | -1.3 [-1.5 to -1.0] | -1.0 [-1.2 to -0.8]
Statistical Analysis 1: Comparison: MK-8189 16 mg vs Placebo and MK-8189 24 mg; Test type: Superiority — It was hypothesized that MK-8189 16 mg is superior to placebo in reducing Week 6 CGI-S change from baseline; p = 0.254, ANCOVA; LS Mean Difference = -0.2, 97.5% CI 2-sided [-0.5 to 0.1]
Statistical Analysis 2: Comparison: MK-8189 24 mg vs Placebo and MK-8189 24 mg; Test type: Superiority — It was hypothesized that MK-8189 24 mg is superior to placebo in reducing Week 6 CGI-S change from baseline; p = 0.959, ANCOVA; LS Mean Difference = 0.0, 97.5% CI 2-sided [-0.3 to 0.3]

5. Secondary Outcome: Change From Baseline in Body Weight at Week 12
Description: The change from baseline in body weigh was determined at Week 12. Negative and positive values represent body weight loss and gain from baseline, respectively. Weight was measured using a standardized scale. Risperidone and placebo were active and inactive controls, respectively.
Time Frame: Baseline and Week 12
Population: All participants who received ≥1 dose of MK-8189, risperidone, or placebo, and have both a baseline measurement and ≥1 valid post-baseline assessment, are included.
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | MK-8189 8 mg | MK-8189 16 mg | MK-8189 24 mg | Risperidone 6 mg | Placebo and MK-8189 24 mg
Number analyzed (Participants) | 12 | 56 | 45 | 34 | 52
Kilograms | -3.2 (5.4) | -5.0 (5.6) | -2.9 (5.1) | 2.7 (3.8) | -2.0 (3.9)

6. Primary Outcome: Number of Participants Who Discontinued From Study Intervention Due to AE
Description: as for outcome 2
Time Frame: Up to Week 6
Population: All participants who received ≥1 dose of study intervention are included.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-8189 8 mg | MK-8189 16 mg | MK-8189 24 mg | Risperidone 6 mg | Placebo and MK-8189 24 mg
Number analyzed (Participants) | 41 | 132 | 132 | 65 | 129
Participants | 8 | 17 | 33 | 8 | 16

7. Secondary Outcome: Change From Baseline in Body Weight at Week 6
Description: The change from baseline in body weigh was determined at Week 6. Negative and positive values represent body weight loss and gain from baseline, respectively. Weight was measured using a standardized scale. Risperidone and placebo were active and inactive controls, respectively.
Time Frame: Baseline and Week 6
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | MK-8189 8 mg | MK-8189 16 mg | MK-8189 24 mg | Risperidone 6 mg | Placebo and MK-8189 24 mg
Number analyzed (Participants) | 19 | 86 | 75 | 44 | 91
Kilograms | -1.1 (3.0) | -3.2 (4.1) | -2.4 (3.8) | 2.6 (3.4) | 0.5 (3.5)

8. Secondary Outcome: Change From Baseline in Body Weight at Week 12: Model-based Analysis
Description: as for outcome 5
Time Frame: Baseline and Week 12
Population: All participants who received ≥1 dose of MK-8189 (16 or 24 mg), risperidone, or placebo, and have both a baseline measurement and ≥1 valid post-baseline assessment, are included. Per protocol, the 8 mg arm was excluded from analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Kilograms
Arm/Group | MK-8189 8 mg | MK-8189 16 mg | MK-8189 24 mg | Risperidone 6 mg | Placebo and MK-8189 24 mg
Number analyzed (Participants) | 0 | 56 | 45 | 34 | 52
Kilograms |  | -5.4 [-6.5 to -4.4] | -4.3 [-5.4 to -3.2] | 3.0 [1.6 to 4.4] | -2.3 [-3.4 to -1.3]
Statistical Analysis 1: Comparison: MK-8189 16 mg vs Risperidone 6 mg; Test type: Superiority — Estimated Treatment Difference vs Risperidone; p < 0.001, ANCOVA; Covariates were treatment, stratum (US Black, US-Non-Black, Other), gender (male, female), and with baseline value, the duration of illness and age; LS Mean Difference = -8.5, 97.5% CI 2-sided [-10.4 to -6.5]
Statistical Analysis 2: Comparison: MK-8189 24 mg vs Risperidone 6 mg; Test type: Superiority — Estimated Treatment Difference vs Risperidone; p < 0.001, ANCOVA; [statistical method as in outcome 8, analysis 1]; LS Mean Difference = -7.3, 97.5% CI 2-sided [-9.3 to -5.2]

9. Secondary Outcome: Change From Baseline in Body Weight at Week 6: Model-based Analysis
Description: as for outcome 7
Time Frame: Baseline and Week 6
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: Kilograms
Arm/Group | MK-8189 8 mg | MK-8189 16 mg | MK-8189 24 mg | Risperidone 6 mg | Placebo and MK-8189 24 mg
Number analyzed (Participants) | 0 | 86 | 75 | 44 | 91
Kilograms |  | -3.2 [-3.9 to -2.5] | -2.8 [-3.5 to -2.1] | 2.8 [1.8 to 3.8] | 0.5 [-0.2 to 1.2]
Statistical Analysis 1: Comparison: MK-8189 16 mg vs Risperidone 6 mg; Test type: Superiority — Estimated Treatment Difference vs Risperidone; p < 0.001, ANCOVA; [statistical method as in outcome 8, analysis 1]; LS Mean Difference = -6.0, 97.5% CI 2-sided [-7.4 to -4.6]
Statistical Analysis 2: Comparison: MK-8189 24 mg vs Risperidone 6 mg; Test type: Superiority — Estimated Treatment Difference vs Risperidone; p < 0.001, ANCOVA; [statistical method as in outcome 8, analysis 1]; LS Mean Difference = -5.6, 97.5% CI 2-sided [-7.0 to -4.2]

ADVERSE EVENTS:
Time Frame: Up to ~14 weeks
Description: All treated participants are included. To accommodate the different treatments in the "Placebo and MK-8189 24 mg", data from Weeks 1 to 6 and Weeks 7 to 12 are presented separately.
Groups:
- MK-8189 8 mg Weeks 1 to 6: Participants received MK-8189 8 mg QD from Weeks 1 to 6.
- MK-8189 16 mg Weeks 1 to 6: Participants (who received MK-8189 16 mg Weeks 1 to 6) received MK-8189 16 mg QD from Weeks 1 to 6.
- MK-8189 24 mg Weeks 1 to 6: Participants received MK-8189 24 mg QD from Weeks 1 to 6.
- Risperidone 6 mg Weeks 1 to 6: Participants received risperidone 6 mg QD from Weeks 1 to 6.
- Placebo Weeks 1 to 6: Participants received placebo QD from Weeks 1 to 6.
- MK-8189 8 mg Weeks 7 to 12: Participants (who received MK-8189 8 mg Weeks 1 to 6) received MK-8189 8 mg QD from Weeks 7 to 12.
- MK-8189 16 mg Weeks 7 to 12: Participants (who received MK-8189 16 mg Weeks 1 to 6) received MK-8189 16 mg QD from Weeks 7 to 12.
- MK-8189 24 mg Weeks 7 to 12: Participants (who received MK-8189 24 mg) received MK-8189 24 mg QD from Weeks 7 to 12.
- Risperidone 6 mg Weeks 7 to 12: Participants (who received risperidone 6 mg Weeks 1 to 6) received risperidone 8 mg QD from Weeks 7 to 12.
- MK-8189 24 mg Weeks 7 to 12 (Placebo Weeks 1 to 6): Participants (who received placebo Weeks 1 to 6) received MK-8189 24 mg Weeks 7 to 12.
Arm/Group | MK-8189 8 mg Weeks 1 to 6 | MK-8189 16 mg Weeks 1 to 6 | MK-8189 24 mg Weeks 1 to 6 | Risperidone 6 mg Weeks 1 to 6 | Placebo Weeks 1 to 6 | MK-8189 8 mg Weeks 7 to 12 | MK-8189 16 mg Weeks 7 to 12 | MK-8189 24 mg Weeks 7 to 12 | Risperidone 6 mg Weeks 7 to 12 | MK-8189 24 mg Weeks 7 to 12 (Placebo Weeks 1 to 6)
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/132 | 0/132 | 0/65 | 0/129 | 0/17 | 1/75 | 0/60 | 0/39 | 0/85
Serious Adverse Events (participants affected / at risk) | 1/41 | 8/132 | 6/132 | 2/65 | 0/129 | 3/17 | 4/75 | 3/60 | 0/39 | 2/85
Other Adverse Events (participants affected / at risk) | 18/41 | 58/132 | 72/132 | 19/65 | 45/129 | 4/17 | 18/75 | 10/60 | 9/39 | 25/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MK-8189 8 mg Weeks 1 to 6 (N=41) | MK-8189 16 mg Weeks 1 to 6 (N=132) | MK-8189 24 mg Weeks 1 to 6 (N=132) | Risperidone 6 mg Weeks 1 to 6 (N=65) | Placebo Weeks 1 to 6 (N=129) | MK-8189 8 mg Weeks 7 to 12 (N=17) | MK-8189 16 mg Weeks 7 to 12 (N=75) | MK-8189 24 mg Weeks 7 to 12 (N=60) | Risperidone 6 mg Weeks 7 to 12 (N=39) | MK-8189 24 mg Weeks 7 to 12 (Placebo Weeks 1 to 6) (N=85)
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Schizophrenia (Psychiatric disorders) | 1 | 2 | 5 | 1 | 0 | 2 | 3 | 2 | 0 | 2
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8189 8 mg Weeks 1 to 6 (N=41) | MK-8189 16 mg Weeks 1 to 6 (N=132) | MK-8189 24 mg Weeks 1 to 6 (N=132) | Risperidone 6 mg Weeks 1 to 6 (N=65) | Placebo Weeks 1 to 6 (N=129) | MK-8189 8 mg Weeks 7 to 12 (N=17) | MK-8189 16 mg Weeks 7 to 12 (N=75) | MK-8189 24 mg Weeks 7 to 12 (N=60) | Risperidone 6 mg Weeks 7 to 12 (N=39) | MK-8189 24 mg Weeks 7 to 12 (Placebo Weeks 1 to 6) (N=85)
Constipation (Gastrointestinal disorders) | 1 (1) | 7 (7) | 3 (4) | 1 (1) | 5 (6) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 6 (6) | 3 (3) | 0 (0) | 5 (5) | 0 (0) | 1 (3) | 1 (1) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2) | 21 (25) | 25 (30) | 6 (11) | 6 (7) | 0 (0) | 3 (6) | 2 (2) | 0 (0) | 5 (5)
Toothache (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 16 (21) | 18 (34) | 1 (4) | 7 (8) | 0 (0) | 4 (5) | 2 (3) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (3) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Akathisia (Nervous system disorders) | 0 (0) | 8 (9) | 12 (12) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (4)
Dystonia (Nervous system disorders) | 2 (2) | 4 (4) | 9 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 12 (12) | 11 (13) | 4 (4) | 12 (12) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 4 (4)
Agitation (Psychiatric disorders) | 4 (5) | 7 (8) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Anxiety (Psychiatric disorders) | 2 (2) | 8 (8) | 13 (13) | 4 (4) | 8 (12) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 4 (5)
Insomnia (Psychiatric disorders) | 4 (4) | 7 (11) | 10 (13) | 1 (1) | 8 (8) | 0 (0) | 7 (7) | 2 (2) | 0 (0) | 4 (4)
Schizophrenia (Psychiatric disorders) | 2 (2) | 6 (6) | 11 (11) | 2 (2) | 7 (7) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 6 (6)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-16): https://cdn.clinicaltrials.gov/large-docs/43/NCT04624243/Prot_SAP_000.pdf